CLINICAL TRIAL: NCT04377555
Title: An Open-Label, Prospective, Single-arm, Multi-center Study to Assess Disease Activity and Biomarkers of Neuronal Damage in Minority Patients With Relapsing Multiple Sclerosis Receiving Treatment With Ocrelizumab
Brief Title: Prospective Study to Assess Disease Activity and Biomarkers in Minority Participants With Relapsing Multiple Sclerosis (RMS) After Initiation and During Treatment With Ocrelizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42071
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis, Relapsing
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Main study participants will be evaluated at baseline, monitored and followed for a 1 year period with the option to participate in a 1 year extension. Participants in the CSF substudy will be followed for two years and will receive two additional doses of 600 mg ocrelizumab at Weeks 48 and 72.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered intravenously (IV) at a dose of 600 mg every 24 weeks. The first dose of ocrelizumab will be administered as two 300 mg IV infusions given 14 days apart. For the subsequent dose, ocrelizumab will be administered as a single 600 mg IV infusion every 24 weeks.

SUMMARY:
Open-label, prospective, single-arm, multi-center study to assess disease activity and biomarker of neuronal damage in minority patients (self-identified Black or African American (AA) and Hispanic/Latino (HA) patients with relapsing multiple sclerosis (RMS) receiving treatment with Ocrelizumab. The study plans to enroll approximately 150 participants (75 AA and 75 HA) with 50 participants enrolled in a CSF sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RMS with Expanded Disability Status Scale (EDSS) 0-5.5 at enrollment
* Participants who self-identify as Black or African American or Hispanic/Latino American
* Treatment-naïve or initiating first or second switch from receiving treatment with certain disease modifying therapies (DMTs) including interferon or glatiramer acetate or dimethyl fumarate (DMF); or siponimod; or fingolimod; or diroximel fumarate; or teriflunomide; or ozanimod; or natalizumab
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for 6 months after the final dose of ocrelizumab
* Neurologically stable for at least 30 days prior to randomization and baseline assessments

Exclusion Criteria:

* Diagnosis of secondary progressive MS without relapses for at least 1 year (nonactive or inactive SPMS)
* Primary Progressive Multiple Sclerosis (PPMS)
* Participants with contraindication to gadolinium based contrast agent for MRI and participants who cannot tolerate MRI procedure
* Infection Related
* Cancer Related
* Pregnant or lactating, or intending to become pregnant during the study
* Other Medical Conditions
* Known presence or history of other neurologic disorders
* Vaccinations: Receipt of a live vaccine, or attenuated, or inactivated / component vaccine within 6 weeks prior to first administration of ocrelizumab
* Laboratory: abnormalities or findings at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Free of Any Protocol-defined Events During a 48-week Period on Treatment | 48 Weeks
  A protocol-defined event is the occurrence of at least one of the following: a protocol-defined relapse; a 24-week Confirmed Disability Progression event; a T1 Gd-enhancing lesion or new and/or enlarging T2 lesion on brain magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Time to onset of 24 weeks confirmed disability progression (CDP) at week 48 | Week 48
Time to protocol-defined event | Week 48
  A protocol-defined event is the occurrence of at least one of the following: a protocol-defined relapse; a 24-week Confirmed Disability Progression event; a T1 Gd-enhancing lesion or new and/or enlarging T2 lesion on brain MRI
Annualized relapse rate at week 48 | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (26):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Keck School of Medicine of USC, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Baptist Neurology - Beaches, Jacksonville Beach, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Shepherd Center Inc., Atlanta, Georgia
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Josephson Wallack Munshower Neurology PC, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University Neurology Research Office, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Paramus, New Jersey
  - SUNY Upstate Medical Center, Syracuse, New York
  - Guilford Neurologic Research Partners, LLC, Greensboro, North Carolina
  - Jefferson University Hospitals, Thomas Jefferson University, Philadelphia, Pennsylvania
  - Neurology Clinic - Cordova, Cordova, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - North Texas Institute of Neurology and Headache NextStage Clinical Research Clinic, Frisco, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Multiple Sclerosis Center of Tidewater, Norfolk, Virginia
  - Wheaton Franciscan Healthcare - St. Francis Outpatient Center, Milwaukee, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- The Aga Khan University-Kenya., Nairobi, Kenya
- Centro Internacional De Mercadeo, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Williams MJ, Okai AF, Cross AH, Monson NL, Vartanian T, Thrower BW, Reder AT, English JB, Wu GF, Bernitsas E, Yap S, Ndrio J, Pei J, Mowry EM, Magrini F, Acosta J, Amezcua L; CHIMES investigators. Demographics and baseline disease characteristics of Black and Hispanic patients with multiple sclerosis in the open-label, single-arm, multicenter, phase IV CHIMES trial. Mult Scler Relat Disord. 2023 Aug;76:104794. doi: 10.1016/j.msard.2023.104794. Epub 2023 Jun 9. PMID 37356256